CLINICAL TRIAL: NCT02895893
Title: PrEP SMART PHASE I TRIAL
Acronym: PrepSmart
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Intelligent Automation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00071752
Record Dates: First submitted 2016-08-30; First posted 2016-09-12 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2016-07

CONDITIONS: At Risk for HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Smartphone app condition (Experimental): Men who are at risk for HIV and already prescribed and taking Truvada will be asked to use an application on their smart phones called "PrEP Smart".
  Interventions: Behavioral: PrEP Smart

INTERVENTIONS:
Behavioral: PrEP Smart — Men who have sex with men and already prescribed and taking oral PrEP will use an application on their smart phone for 4 weeks.

SUMMARY:
The goal of this Phase I study is to conduct a proof-of-concept trial of a contingency management (CM) targeting adherence to oral HIV antiretroviral pre-exposure prophylaxis (PrEP) administered via a smartphone-based medication adherence platform (PrEP SMART, "the app").

DETAILED DESCRIPTION:
The goal of this Phase I study is to conduct a proof-of-concept trial of a contingency management (CM) targeting adherence to oral HIV antiretroviral pre-exposure prophylaxis (PrEP) administered via a smartphone-based medication adherence platform (PrEP SMART, "the app").

PrEP provides a strong preventative benefit to individuals at-risk for HIV. While oral PrEP adherence is highly correlated with its efficacy in clinical trials, adherence rates are variable and range from 29-80%. In real-world practice settings, PrEP adherence may even be lower. As such, interventions are needed to improve and sustain adherence to oral PrEP, thereby maximizing preventative benefits in at-risk populations.

CM is a behavioral intervention that involves the systematic use of reinforcement dependent on the occurrence of a predefined behavior. CM improves adherence to antiretroviral therapy and post-exposure prophylaxis, but CM has yet to be applied to PrEP adherence. The investigative team recently developed a smartphone-based platform for medication adherence that can integrate CM. Given that mobile technologies such as smartphones are increasingly ubiquitous, a CM-based program administered via smartphone may be a practical intervention that augments PrEP adherence.

In the proposed research, PrEP SMART will provide medication reminders; monetary incentives for daily, verified adherence to PrEP; education about oral PrEP; and assess potential adherence barriers. This will be a 4-week open-label, stage I trial in a community sample of young men who have sex with men (YMSM, n = 12) already prescribed and taking oral PrEP (ages 18-30). YMSM were selected because they are the only high risk group experiencing an increase in HIV incidence in the U.S.

The investigative team is particularly well-positioned as we have expertise in the development of mobile apps to improve medication adherence, including in the context of HIV care; oral PrEP efficacy trials; and are conducting research using the "parent version" of PrEP SMART (mSMART; Mobile App based Personalized Solutions and Tools for Medication Adherence of Rx Pill) platform in another clinical context.

The primary aim of this study is to conduct a proof-of-concept trial of PrEP SMART.

* Aim 1a: User interaction with the app will allow for evaluation of feasibility (e.g., the number of app uses/day)
* Aim 1b: Acceptability will be assessed via self-report ratings and qualitative interviewing
* Aim 1c: Medication adherence will be evaluated via daily smartphone camera-based medication event assessments to establish preliminary data on the impact of mSMART for future efficacy trials.
* Aim 1d: Adherence barriers will be evaluated by mSMART following missed doses.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-30 years of age
* Self-report having sex with men in the past 6 months
* Currently prescribed PrEP (Truvada) for HIV prevention
* English-speaking
* Participant has an Android or iOS smartphone

Exclusion Criteria:

* History of chronic/significant medical or psychiatric condition that will interfere with study participation
* Unable to attend sessions

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07; Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by the average number of times per day participants initiate an interaction with PrEP Smart | 4 weeks
Feasibility as measured by the average number of times per day subjects respond to a prompt from PrEP Smart over the course of the four week period. | 4 weeks

SECONDARY OUTCOMES:
Barriers to adherence following missed doses as measured by daily PrEP Smart assessment. | 4 weeks
Acceptability as measured by questionnaire that includes questions about satisfaction and likelihood of recommending to others on a Likert scale of 1 to 4. | 4 weeks
Acceptability as measured by an interview that will be conducted by the Principal Investigator. | 4 weeks
Barriers to adherence will be measured by the number of times it was taken outside of a 1 hour window | 4 weeks
Barriers to adherence will be measured by self-report via the PrEP Smart application. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Mitchell, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mitchell JT, LeGrand S, Hightow-Weidman LB, McKellar MS, Kashuba AD, Cottrell M, McLaurin T, Satapathy G, McClernon FJ. Smartphone-Based Contingency Management Intervention to Improve Pre-Exposure Prophylaxis Adherence: Pilot Trial. JMIR Mhealth Uhealth. 2018 Sep 10;6(9):e10456. doi: 10.2196/10456. PMID 30201601